CLINICAL TRIAL: NCT05320679
Title: Development and Implementation of Pain Related Avoidance of Movement
Brief Title: Development of Pain Related Avoidance of Movement Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Yavuz Yakut, Professor, Hasan Kalyoncu University
Other Study IDs: 2020/021
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Musculoskeletal Pain; Low Back Pain; Back Pain
Keywords: Musculoskeletal pain; Kinesiophobia; Questionnaire
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain; Back Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients who have musculoskeletal pain
  Interventions: Other: Implementation of Questionnaire

INTERVENTIONS:
Other: Implementation of Questionnaire — Compartment of results of questionnaires which already been used in literature and results of developing Pain Related Avoidance of Movement Questionnaire

SUMMARY:
In recent studies, it has been shown that people may have avoidance of movement due to pain. However, there is no scale that evaluates avoidance of movement due to pain in musculoskeletal problems. The aim of this study is to develop a scale to measure how much pain-related movement and activity is avoided in individuals with musculoskeletal pain, and to examine the results of its clinical application.

DETAILED DESCRIPTION:
Approaches and methods to be applied in the research;

* Demographic information (age, gender, weight, height, pain location, pain duration and diagnose) form will be recorded.
* Creation of questionnaire items
* Reviewing of items/questions
* Patients who accept to fill out the questionnaire and who has complain of musculoskeletal pain will be asked to answer the questions.
* Editing the scale according to the answers
* Reliability and validity studies of the questionnaire
* Investigation of the results of applying the scale with clinical follow-up

To compare results of Pain-Related Avoidance of Movement Questionnaire following common used questionnaires are going to be used;

* Visual Analogue Scale (VAS)
* Tampa Kinesiophobia Scale
* Oswestry Low Back Pain and Disability Index-2.0

SPSS version 23 (SPSS Inc, Armonk, NY) program will be used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria;

* Having agreed to fill out the questionnaire
* Having pain caused by problems related to the musculoskeletal system
* Not having any disability in performing activities of daily living

Exclusion Criteria;

* Individuals who are not allowed to move due to pain
* If they have undergone surgery, individuals who have inconveniences in moving due to surgery
* Individuals who have cognitive problems in completing the questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are going to be patients who have musculoskeletal pain problem.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Total points of Pain Related Avoidance of Movement Questionnaire | 1 week
  Pain related avoidance of movement score is going to be assess by Pain Related Avoidance of Movement Questionnaire to determine change from baseline and, to examine correlation of other questionnaires.

SECONDARY OUTCOMES:
Change from baseline score in pain score | 1 week
  Pain score is going to be assess by VAS to determine change from baseline. Normal range of VAS score is between 0 point to 10 points. Higher score means worse pain level.
Change from baseline score in kinesiophobia score | 1 week
  Kinesiophobia score is going to be assess by Tampa Kinesiophobia Scale to determine change from baseline. The normal range of kinesiophobia score is between 17 points to 68 points. Higher score means worse kinesiophobia level.
Change from baseline in disability score | 1 week
  Disability score is going to be assess by Oswestry Disability Index to determine the change from baseline. The normal range of percentage is between 0 to 100. Higher percentage means worse disability level.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)